CLINICAL TRIAL: NCT02675309
Title: A Study to Investigate the Effect of MT-8554 on the Pharmacokinetics of Simvastatin and Rosuvastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MT-8554-E05
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MT-8554, rosuvastatin and simvastatin (Experimental): Subjects will be administered a single dose of rosuvastatin followed on Day 4 by a single dose of simvastatin. MT-8554 will be administered from Days 6 to 12 with co-administration of rosuvastatin and simvastatin on Days 9 and 12, respectively.
  Interventions: Drug: MT-8554; Drug: rosuvastatin; Drug: simvastatin

INTERVENTIONS:
Drug: MT-8554
Drug: rosuvastatin
Drug: simvastatin

SUMMARY:
The purpose of this study is to investigate the effect of MT-8554 on the pharmacokinetics of simvastatin and rosuvastatin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free from clinically significant illness or disease
* Male Caucasian subjects aged 18 to 55
* A body weight of ≥60 kg

Exclusion Criteria:

* Participation in more than three clinical studies involving administration of an Investigational Medicinal Product in the previous year, or any study within 12 weeks.
* Clinically significant endocrine, thyroid, hepatic, respiratory, gastro-intestinal, renal, cardiovascular disease, or history of any significant psychiatric/psychotic illness disorder.
* Clinically relevant abnormal medical history, physical findings or laboratory values

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of rosuvastatin alone and in the presence of MT-8554. | 72 hours post dose
Cmax of rosuvastatin alone and in the presence of MT-8554. | 72 hours post dose
AUC of simvastatin/simvastatin acid alone and in the presence of MT-8554. | 24 hours post dose
Cmax of simvastatin/simvastatin acid alone and in the presence of MT-8554. | 24 hours post dose

SECONDARY OUTCOMES:
Safety and Tolerability as measured by vital signs | Up to Day 16
Safety and Tolerability as measured by number of participants with adverse events | Up to Day 16

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational center, City Name, United Kingdom